CLINICAL TRIAL: NCT02777580
Title: STrategic Reperfusion in Elderly Patients Early After Myocardial Infarction
Acronym: STREAM-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Boehringer Ingelheim (Industry); Life Sciences Research Partners (Other); Frans Van de Werf Fund for Clinical Cardiovascular Research (Other)
Responsible Party: Principal Investigator, Frans Van de Werf, Prof Dr, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LRD.2016.STREAM2
Record Dates: First submitted 2016-05-13; First posted 2016-05-19 (Estimated); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-07

CONDITIONS: Myocardial Infarction
Keywords: Thrombolytic Therapy; Primary PCI
MeSH Terms: conditions — Myocardial Infarction | interventions — Tenecteplase; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmaco-invasive strategy (Experimental): Half-dose tenecteplase and additional antiplatelet therapy with a loading dose of 300 mg clopidogrel, aspirin and coupled with antithrombin therapy followed by coronary angiography within 6-24 hours or rescue coronary intervention as required.
  Interventions: Drug: Tenecteplase; Drug: Clopidogrel; Procedure: Coronary angiography
- Standard primary PCI (Active Comparator): Primary PCI with a P2Y12 antagonist and antithrombin treatment according to local standards.
  Interventions: Procedure: Primary PCI

INTERVENTIONS:
Drug: Tenecteplase — Half dose Tenecteplase
  Other Names: TNKase; Metalyse
  Arms: Pharmaco-invasive strategy
Drug: Clopidogrel — 300 mg p.o. initial loading dose. Maintenance dose of 75 mg p.o. once daily. The maintenance dose of Clopidogrel (75 mg p.o. per day) should be continued for 1 year.
  Arms: Pharmaco-invasive strategy
Procedure: Coronary angiography — Coronary angiography followed by PCI or CABG if required, rescue PCI if required
  Arms: Pharmaco-invasive strategy
Procedure: Primary PCI — Primary PCI accoring to local standards
  Arms: Standard primary PCI

SUMMARY:
In patients ≥ 60yrs with acute ST-elevation myocardial infarction randomised within 3 hours of onset of symptoms the efficacy and safety of a strategy of early fibrinolytic treatment with half-dose tenecteplase and additional antiplatelet therapy with a loading dose of 300 mg clopidogrel, aspirin and coupled with antithrombin therapy followed by catheterisation within 6-24 hours or rescue coronary intervention as required, will be compared to a strategy of primary PCI with a P2Y12 antagonist and antithrombin treatment according to local standards.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal or greater than 60 years
2. Onset of symptoms < 3 hours prior to randomisation
3. 12-lead ECG indicative of an acute STEMI (ST-elevation will be measured from the J point; scale: 1 mm per 0.1 mV):

   * ≥ 2 mm ST-elevation across 2 contiguous precordial leads (V1-V6) or leads I and aVL for a minimum combined total of ≥ 4 mm ST-elevation or
   * ≥ 2 mm ST-elevation in 2 contiguous inferior leads (II, III, aVF) for a minimum combined total of ≥ 4 mm ST-elevation
4. Informed consent received

Exclusion Criteria:

1. 1. Expected performance of PCI < 60 minutes from diagnosis (qualifying ECG) or inability to arrive at the catheterisation laboratory within 3 hours
2. Previous CABG
3. Left bundle branch block or ventricular pacing
4. Patients with cardiogenic shock - Killip Class 4
5. Patients with a body weight < 55 kg (known or estimated)
6. Uncontrolled hypertension, defined as sustained blood pressure ≥ 180/110 mm Hg (systolic BP ≥ 180 mm Hg and/or diastolic BP ≥ 110 mm Hg) prior to randomisation
7. Known prior stroke or TIA
8. Recent administration of any i.v. or s.c. anticoagulation within 12 hours, including unfractionated heparin, enoxaparin, and/or bivalirudin or current use of oral anticoagulation (i.e. warfarin or a NOACs)
9. Active bleeding or known bleeding disorder/diathesis
10. Known history of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery) or recent trauma to the head or cranium (i.e. < 3 months)
11. Major surgery, biopsy of a parenchymal organ, or significant trauma within the past 2 months (this includes any trauma associated with the current myocardial infarction)
12. Clinical diagnosis associated with increased risk of bleeding including known active peptic ulceration and/or neoplasm with increased bleeding risk
13. Prolonged cardiopulmonary resuscitation (> 2 minutes) within the past 2 weeks
14. Known acute pericarditis and/or subacute bacterial endocarditis
15. Known acute pancreatitis or known severe hepatic dysfunction, including hepatic failure, cirrhosis, portal hypertension (oesophageal varices) and active hepatitis
16. Dementia
17. Known severe renal insufficiency
18. Previous enrolment in this study or treatment with an investigational drug or device under another study protocol in the past 7 days
19. Known allergic reactions to tenecteplase, clopidogrel, enoxaparin and aspirin
20. Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk if the investigational therapy is initiated.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frans Van de Werf, MD, PhD, Study Chair — KU Leuven; Paul Armstrong, MD, Study Chair — University of Alberta, Edmonton, Canada; Peter Sinnaeve, MD, PhD, Principal Investigator — UZ Leuven, Belgium; Robert Welsh, MD, Principal Investigator — University of Alberta, Edmonton, Canada; Patrick Goldstein, MD, Principal Investigator — Lille University Hospital, France
Locations (50):
- Liverpool Hospital - Cardiology Department, Liverpool, Australia
- Centro de Pesquisa São Lucas - Hospital E Maternidade Celso Pierro, Campinas, Brazil
- University of Alberta Hospital, Edmonton, Alberta, Canada
- Chile (8):
  - Hospital Regional de Antofagasta, Antofagasta
  - Hospital Comunitario de Mejillones, Mejillones
  - Hospital de Melipilla, Melipilla
  - Hospital Regional de Rancagua, Rancagua
  - SAR Rancagua, Rancagua
  - Hospital San Juan de Dios, Santiago
  - Hospital de Talagante, Talagante
  - Hospital de Tocopilla, Tocopilla
- France (11):
  - CH Louis Pradel - Hospices civils de Lyon, Bron
  - CH Cahors - SAMU 46, Cahors
  - CH de Chateauroux, Châteauroux
  - CH Sud Francilien - Service Cardiologie, Corbeil-Essonnes
  - Centre Hospitalier de Versailles, Le Chesnay
  - CHRU de Lille, Lille
  - CH St. Joseph - St Luc - Lyon, Lyon
  - Groupe Hospitalier Sud Ile de France - CH de Melun - Service SAMU 77, Melun
  - Clinque du Pont de Chaume, Montauban
  - CHU de Rennes, Rennes
  - CH Lucien Hussel, Vienne
- Mexico (2):
  - Hospital Gea Gonzalez, Mexico City
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City
- Montenegro (4):
  - JZU Blazo Orlandic, Bar
  - General Hospital Danilo the First Cetinje, Cetinje
  - General Hospital of Niksic, Nikšić
  - Clinical Centar of Montenegro, Podgorica
- Russia (6):
  - Federal State Budgetary Inst "Research Inst. for Complex Issues of Card. Diseases", Kemerovo
  - State Budgetary Healthcare Inst. Kemerovo-Clinical Emergency Care Station, Kemerovo
  - Federal State Budgetary Scientific Inst "Tomsk Nat Research Med.Center of Russian Academy Sciences", Tomsk
  - Tomsk Regional State Autonomous Healthcare Institution Emergency Care Station, Tomsk
  - State Budgetary Healthcare Institution of Tverskoy Region "Region Clinical Hospital", Tver'
  - Tver Region State Budgetary Healthcare Institution "Tver Emergency Station", Tver'
- Serbia (12):
  - Clinical Center of Serbia, Cardiology Clinic, Belgrade
  - Military Medical Academy, Clinic for Emergency Internal Medicine, Belgrade
  - Institute for cardiovascular diseases Dedinje, Cardiovascular research sector, Belgrade
  - General Hospital Cuprija, Cardiology Department, Ćuprija
  - General Hospital Jagodina/Intenal Medicine department, Jagodina
  - Institute for cardiovascular diseases Vojvodina - Sremska Kamenica, Cardiology Clinic, Kamenitz
  - Clinical Center Kragujevac, Cardiology Clinic, Kragujevac
  - General Hospital Pancevo/Department of internal medicine - cardiology section, Pančevo
  - General Hospital "Sveti Luka" Smederevo, Dept of Internal Med - Cardiology Section, Smederevo
  - General Hospital "Dr. Laza K. Lazarevic" Sabac, Internal medicine department, Šabac
  - Opsta bolnica Vrbas, Cardiology Department, Vrbas
  - General Hospital Vrsac/Cardiology department with coronary unit, Vršac
- Spain (4):
  - Hospital Virgen de la Victoria, Unidad de Cuidados Intensivos, Málaga
  - Hospital de Antequera, Unidad de Cuidados Intensivos, Málaga
  - Hospital Serrania Ronda, Unidad de Cuidados Intensivos, Málaga
  - Hospital Comarcal Axarquia, Unidad de Cuidados Intensivos, Málaga

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Armstrong PW, Gershlick AH, Goldstein P, Wilcox R, Danays T, Lambert Y, Sulimov V, Rosell Ortiz F, Ostojic M, Welsh RC, Carvalho AC, Nanas J, Arntz HR, Halvorsen S, Huber K, Grajek S, Fresco C, Bluhmki E, Regelin A, Vandenberghe K, Bogaerts K, Van de Werf F; STREAM Investigative Team. Fibrinolysis or primary PCI in ST-segment elevation myocardial infarction. N Engl J Med. 2013 Apr 11;368(15):1379-87. doi: 10.1056/NEJMoa1301092. Epub 2013 Mar 10. PMID 23473396
- [Background] Sinnaeve PR, Armstrong PW, Gershlick AH, Goldstein P, Wilcox R, Lambert Y, Danays T, Soulat L, Halvorsen S, Ortiz FR, Vandenberghe K, Regelin A, Bluhmki E, Bogaerts K, Van de Werf F; STREAM investigators. ST-segment-elevation myocardial infarction patients randomized to a pharmaco-invasive strategy or primary percutaneous coronary intervention: Strategic Reperfusion Early After Myocardial Infarction (STREAM) 1-year mortality follow-up. Circulation. 2014 Sep 30;130(14):1139-45. doi: 10.1161/CIRCULATIONAHA.114.009570. Epub 2014 Aug 26. PMID 25161043
- [Background] Dianati Maleki N, Van de Werf F, Goldstein P, Adgey JA, Lambert Y, Sulimov V, Rosell-Ortiz F, Gershlick AH, Zheng Y, Westerhout CM, Armstrong PW. Aborted myocardial infarction in ST-elevation myocardial infarction: insights from the STrategic Reperfusion Early After Myocardial infarction trial. Heart. 2014 Oct;100(19):1543-9. doi: 10.1136/heartjnl-2014-306023. Epub 2014 Jun 10. PMID 24916050
- [Background] Sinnaeve PR, Danays T, Bogaerts K, Van de Werf F, Armstrong PW. Drug Treatment of STEMI in the Elderly: Focus on Fibrinolytic Therapy and Insights from the STREAM Trial. Drugs Aging. 2016 Feb;33(2):109-18. doi: 10.1007/s40266-016-0345-6. PMID 26849132
- [Derived] Armstrong PW, Zheng Y, Welsh RC, Sinnaeve PR, de Werf FV, Westerhout CM, Bainey KR. Primary Percutaneous Coronary Intervention within the First Hour: Insights from Early-Treated Patients with ST-Elevation Myocardial Infarction. Am Heart J. 2026 Jan 29:107363. doi: 10.1016/j.ahj.2026.107363. Online ahead of print. PMID 41619999
- [Derived] Bainey KR, Welsh RC, Zheng Y, Arias-Mendoza A, Ristic AD, Averkov OV, Lambert Y, Temple T, Ly E, Bogaerts K, Sinnaeve P, Westerhout CM, Van de Werf F, Armstrong PW; STREAM-2 Investigators. Pharmaco-invasive strategy and dosing of tenecteplase in STEMI patients 60 to <75 years: An inter-trial comparison of the STREAM-1 and STREAM-2 trials. Am Heart J. 2025 Jun;284:20-31. doi: 10.1016/j.ahj.2025.02.002. Epub 2025 Feb 12. PMID 39952376
- [Derived] Bainey KR, Welsh RC, Zheng Y, Arias-Mendoza A, Ristic AD, Averkov OV, Lambert Y, Kerr Saraiva JF, Sepulveda P, Rosell-Ortiz F, French JK, Music LB, Temple T, Ly E, Bogaerts K, Sinnaeve PR, Danays T, Westerhout CM, Van de Werf F, Armstrong PW; STREAM-2 Investigators. Pharmaco-Invasive Strategy With Half-Dose Tenecteplase in Patients With STEMI: Prespecified Pooled Analysis of Patients Aged >/=75 Years in STREAM-1 and 2. Circ Cardiovasc Interv. 2024 Dec;17(12):e014251. doi: 10.1161/CIRCINTERVENTIONS.124.014251. Epub 2024 Dec 17. PMID 39689189
- [Derived] Van de Werf F, Ristic AD, Averkov OV, Arias-Mendoza A, Lambert Y, Kerr Saraiva JF, Sepulveda P, Rosell-Ortiz F, French JK, Music LB, Vandenberghe K, Bogaerts K, Westerhout CM, Pages A, Danays T, Bainey KR, Sinnaeve P, Goldstein P, Welsh RC, Armstrong PW; STREAM-2 Investigators. STREAM-2: Half-Dose Tenecteplase or Primary Percutaneous Coronary Intervention in Older Patients With ST-Segment-Elevation Myocardial Infarction: A Randomized, Open-Label Trial. Circulation. 2023 Aug 29;148(9):753-764. doi: 10.1161/CIRCULATIONAHA.123.064521. Epub 2023 Jul 13. PMID 37439219

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pharmaco-invasive Strategy | Standard Primary PCI
Started | 405 | 204
Completed | 401 | 203
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pharmaco-invasive Strategy | Standard Primary PCI | Total
Number analyzed (Participants) | 401 | 203 | 604
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 113 | 47 | 160
  >=65 years | 288 | 156 | 444
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (8) | 71 (8) | 70 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 66 | 197
  Male | 270 | 137 | 407
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 66 | 34 | 100
  Brazil | 14 | 6 | 20
  Mexico | 53 | 28 | 81
  Australia | 6 | 3 | 9
  Chile | 10 | 5 | 15
  France | 28 | 14 | 42
  Serbia | 117 | 60 | 177
  Montenegro | 5 | 3 | 8
  Russia | 95 | 47 | 142
  Spain | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Successful Reperfusion
Description: Worst-lead ST-segment elevation resolution ≥ 50% 30 min post angiogram/PCI
Time Frame: 30 min post angiogram/PCI
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmaco-invasive Strategy | Standard Primary PCI
Number analyzed (Participants) | 358 | 190
Participants | 305 | 149
Statistical Analysis 1: Comparison: Pharmaco-invasive Strategy vs Standard Primary PCI; Test type: Other; p = 0.05, Chi-squared

2. Primary Outcome: Composite Clinical Efficacy End Point: All Cause Death, Shock, CHF and Reinfarction at 30 Days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmaco-invasive Strategy | Standard Primary PCI
Number analyzed (Participants) | 401 | 203
Participants | 51 | 27
Statistical Analysis 1: Comparison: Pharmaco-invasive Strategy vs Standard Primary PCI; Test type: Other; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.62 to 1.48]

3. Primary Outcome: Total Stroke
Description: Number of patients with stroke (intracranial haemorrhage, ischaemic, haemorrhagic conversion)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmaco-invasive Strategy | Standard Primary PCI
Number analyzed (Participants) | 400 | 203
Participants | 9 | 1
Statistical Analysis 1: Comparison: Pharmaco-invasive Strategy vs Standard Primary PCI; Test type: Other; Risk Ratio (RR) = 4.57, 95% CI 2-sided [0.58 to 35.8]

4. Primary Outcome: Major Non-intrancranial Bleedings
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmaco-invasive Strategy | Standard Primary PCI
Number analyzed (Participants) | 401 | 203
Participants | 5 | 2
Statistical Analysis 1: Comparison: Pharmaco-invasive Strategy vs Standard Primary PCI; Test type: Other; Risk Ratio (RR) = 1.27, 95% CI 2-sided [0.25 to 6.48]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Pharmaco-invasive Strategy | Standard Primary PCI
All-Cause Mortality (participants affected / at risk) | 37/401 | 18/203
Serious Adverse Events (participants affected / at risk) | 69/401 | 32/203
Other Adverse Events (participants affected / at risk) | 0/401 | 0/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Pharmaco-invasive Strategy (N=401) | Standard Primary PCI (N=203)
cardiogenic shock (Cardiac disorders) | 18/400 | 11
heart failure (Cardiac disorders) | 14/400 | 9
reinfarction (Cardiac disorders) | 10/400 | 5
intracranial hemorrhage (Nervous system disorders) | 6/400 | 0
ischemic stroke (Nervous system disorders) | 3/400 | 1
major nonintracranial bleeding (Vascular disorders) | 5/400 | 2
acute ventricle septum defect (Cardiac disorders) | 3 | 0
coronary arterial dissection (Cardiac disorders) | 0 | 2
atrial fibrillation (Cardiac disorders) | 3 | 2
Bradycardia (Cardiac disorders) | 1 | 0
cardiac arrest (Cardiac disorders) | 1 | 2
cardiac failure (Cardiac disorders) | 1 | 0
myocardial rupture (Cardiac disorders) | 7 | 1
pericardial effusion (Cardiac disorders) | 0 | 1
pulseless electrical activity (Cardiac disorders) | 1 | 2
sudden death (Cardiac disorders) | 1 | 0
ventricle rupture (Cardiac disorders) | 1 | 0
ventricular asystole (Cardiac disorders) | 0 | 1
ventricular tachycardia (Cardiac disorders) | 4 | 0
ventricular fibrillation (Cardiac disorders) | 4 | 0
Chest pain (Cardiac disorders) | 1 | 0
right venticular failure (Cardiac disorders) | 0 | 1
Death (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Vascular stent thrombosis (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 4 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumotorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT02777580/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT02777580/SAP_001.pdf